CLINICAL TRIAL: NCT04381065
Title: Utilization of Target Ranges to Treat Persons With Parkinson's Disease by Objective Measurement Using the Personal KinetiGraph® (PKG®) Compared to Standard of Care Assessment (TARGET-PwP)- A Randomized Controlled Trial
Brief Title: Utilization of Target Ranges to Treat Persons With Parkinson's Disease by Objective Measurement Using the PKG
Acronym: TARGET-PwP
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Business decision
Sponsor: Global Kinetics Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: Study 004
Record Dates: First submitted 2020-05-01; First posted 2020-05-08 (Actual); Last update posted 2021-02-01 (Actual); Status verified 2021-01

CONDITIONS: Parkinson Disease
Keywords: Personal KinetiGraph® (PKG®) System; Objective Measurement
MeSH Terms: conditions — Parkinson Disease | interventions — Drug Delivery Systems

STUDY DESIGN:
Intervention Model Description: Eligible subjects will be randomized using the Electronic Data Capture (EDC) system in a 1:1 ratio to the PKG- Group (standard of care clinical assessments without use of PKG data) or the PKG+ Group (standard of care clinical assessments plus use of PKG data).
Who Masked: Participant
Masking Description: Subjects will remain blinded to treatment group throughout the life of the trial. Investigator and research staff will be unblinded to the treatment group as they will or will not have access to the PKG data to be incorporated into their standard of care practice.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- PKG+ Group (Experimental): For subjects in the PKG+ Group, participants will wear the PKG watch prior to all study visits in which the study investigator will review and report on the PKG prior to the visit and use the information to guide the discussion with the subject during the clinical assessment.The PKG will be used to determine if the subject is in the target range or out of the target range based on scores provided by the PKG.
  Interventions: Device: Personal KinetiGraph® (PKG®) System
- PKG- Group (Placebo Comparator): For subjects in the PKG- Group, participants will wear the PKG watch prior to all study visits, however the investigator will not have access to the PKG report and will use standard of care to determine clinical treatment plans.
  Interventions: Device: Personal KinetiGraph® (PKG®) Watch

INTERVENTIONS:
Device: Personal KinetiGraph® (PKG®) System — The Personal KinetiGraph (PKG®) System consists of the following:
  * A wrist-worn movement recording device known as the PKG® Watch, designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period
  * Proprietary algorithms to translate raw movement data collected by the PKG® Watch
  * Data-driven report known as the PKG®
  The PKG® provides continuous, objective, ambulatory assessment of the treatable and disabling symptoms of Parkinson's disease including tremor, bradykinesia and dyskinesia. The PKG® also provides an assessment of daytime somnolence and an indication of propensity for impulsive behaviors.
  Arms: PKG+ Group
Device: Personal KinetiGraph® (PKG®) Watch — The Personal KinetiGraph (PKG®) System consists of the following:
  * A wrist-worn movement recording device known as the PKG® Watch, designed to acquire data on the kinematics of movement disorder symptoms over a 6-10 day period
  * Proprietary algorithms to translate raw movement data collected by the PKG® Watch
  Arms: PKG- Group

SUMMARY:
The main objective of this study is to evaluate whether persons with Parkinson's disease (PwP) whose Parkinson's disease (PD) symptoms are uncontrolled have improved clinical patient outcomes and quality of life when managed with the aid of objective measurement and use of PKG target ranges compared to PwP treated using only standard of care (SOC) (medical history, physical examination).

DETAILED DESCRIPTION:
This is a randomized controlled trial (RCT) to compare the value of the Personal KinetiGraph® (PKG®) System and SOC vs. the SOC alone for treatment of PwP. The study aims to evaluate clinical outcomes, quality of life outcomes, health economic benefits, duration of controlled status, and need for additional PD treatment through 3 years follow-up of PwP specifically treated to a target range when using the PKG data in the clinical management of PD in routine clinical care compared to those managed with SOC alone. All subjects will be treated by Movement Disorder Specialists and General Neurologists with expertise in PD. Both groups will be recommended to undergo treatment changes until they reach a "controlled state" that is determined by either the clinician using SOC (PKG- Group) or using recommended target ranges for PKG scores and SOC assessments (PKG+ Group). Investigators will utilize standard available treatments to manage these PwP in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to sign a written informed consent for study participation and comply with all required follow-up visits
* Presumed to have levodopa responsive PD
* Taking levodopa for at least 30 days prior to screening visit
* Planning to continue using levodopa for PD throughout study participation
* Able to increase levodopa by a minimum of 100mg/day
* Age inclusive at the time of consent of 55-80 years
* Has not received a PKG in the last 12 months

Exclusion Criteria:

* Evidence of atypical or secondary parkinsonism
* Presence of any non-parkinsonian tremors
* Contraindication to increasing levodopa
* Requires the addition of or dose adjustment of an anti-dyskinesia medication within the next 4 months
* Those who have received advanced therapies including individuals no longer actively utilizing these therapies, or planning to receive advanced therapies in the next 6 months
* MoCA score <23 at screening visit
* Bedridden, wheelchair confined, or requires the regular use of an assistive gait device
* Predominant sleep period is during the daytime hours of 9am to 6pm (e.g. third shift worker)
* In the investigator's or sponsor's opinion, subject has any unstable or clinically significant condition that would impair the participant's ability to comply with study requirements or interfere with interpretation of the study endpoints

Ages: 55 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-06 (Estimated); Primary Completion 2022-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Change in Patient Outcomes using Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) | 4 months
  The change in MDS-UPDRS Total score at 4 months from baseline defined as sections I, II, III (per core lab measurement) and IV in PwP. The endpoint will be compared between subjects out of target at baseline for those who are treated with SOC and PKG data (PKG+ Group) versus those who are treated per SOC alone (PKG- Group).

SECONDARY OUTCOMES:
Responder rate for total MDS-UPDRS | 4 months
  Percent "responders" for total MDS-UPDRS based on a minimal clinically important change of >4 points (Shulman LM, Gruber-Baldini AL, Anderson KE, et al. The Clinically Important Difference on the Unified Parkinson's Disease Rating Scale. Arch Neurol 2010: 67(1):64-70.). The Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Parts I and II (non-motor) each contain 13 questions/evaluations, Part III (motor) contains 33 and Part IV (motor) contains 6. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Responder rate for PKG | 4 months
  Percent "responders" by PKG (defined as BKS change of >2 point improvement)
Change in MDS-UPDRS motor endpoints | 4 months, 1 year, 2 years, 3 years
  Change in MDS-UPDRS Part III (per core lab measurement). The Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Part III is the motor examination and contains 33 questions/evaluations. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Change in MDS-UPDRS total | 1 year, 2 years, 3 years
  Change in MDS-UPDRS Total score from baseline. The Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Parts I and II (non-motor) each contain 13 questions/evaluations, Part III (motor) contains 33 and Part IV (motor) contains 6. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Change in MDS-UPDRS sub parts | 4 months, 1 year, 2 years, 3 years
  Change in the non-motor (parts I and II) score and change in Part IV for the MDS-UPDRS from baseline. The Movement Disorder Specialist - Unified Parkinson's Disease Rating Scale (MDS-UPDRS) evaluates motor and non-motor symptoms in persons with Parkinson's and consists of 4 parts with various questions and evaluations. Parts I and II (non-motor) each contain 13 questions/evaluations, Part III (motor) contains 33 and Part IV (motor) contains 6. Each question/evaluation score ranges from 0 (normal) to 4 (severe). Higher scores indicate a greater impact of Parkinson's disease symptoms (i.e., worse symptoms).
Change in PKG Bradykinesia Score (BKS) | 4 months, 1 year, 2 years, 3 years
  Change in the PKG reported BKS from baseline. A higher score represents more severe bradykinesia.
Change in PKG Dyskinesia score (DKS) | 4 months, 1 year, 2 years, 3 years
  Change in the PKG reported DKS from baseline. A higher score represents more severe dyskinesia.
Change in Percent Time in Tremor (PTT) | 4 months, 1 year, 2 years, 3 years
  Change in the PKG reported PTT from baseline, max 100%. A PTT of >1% indicates that tremor is present.
Change in Fluctuation Dyskinesia score (FDS) | 4 months, 1 year, 2 years, 3 years
  Change in the PKG reported FDS from baseline. The higher the score, the more severe the fluctuation, and a FDS of 7.5-13 indicates controlled fluctuations.
Change in Percent Time Immobile (PTI) | 4 months, 1 year, 2 years, 3 years
  Change in the PKG reported PTI from baseline, max 100%. A PTI of >5% is considered high.
Change in Parkinson's Disease Questionnaire-39 questions (PDQ-39) | 4 months, 1 year, 2 years, 3 years
  Change in the patient reported quality of life questionnaire PDQ-39 from baseline. The PDQ-39 is a 39-item self-report questionnaire, which assesses Parkinson's disease-specific health related quality of life issues across 8 dimensions. Each dimension total score range from 0 (never have difficulty) to 100 (always have difficulty). Lower scores reflect better quality of life.
Number of Interim Visits | 4 months
  Number of interim visits conducted from baseline to 4 months in each arm

OTHER OUTCOMES:
Levodopa Equivalent Dose (LED) | 4 months, 1 year, 2 years, 3 years
  Levodopa Equivalent Dose (LED) at each visit
PKG Patient Survey | 4 months, 1 year, 2 years, 3 years
  Analyze PKG usability with the PKG Patient reported survey. Questions are on a scale of strongly agree to strongly disagree and will be patient reported information related to their use of the PKG watch. Both treatment groups will be administered the survey and scores will be aggregated by group and compared.
Healthcare Utilization | 4 months, 1 year, 2 years, 3 years
  Rate of protocol defined adverse events affecting health care utilization from baseline
Potential Contraindications | 4 months, 1 year, 2 years, 3 years
  Rate of protocol defined adverse events and potential contraindications for increasing dopaminergic therapy from baseline
Lifestyle Factors Impacted by PD | 4 months, 1 year, 2 years, 3 years
  Rate of protocol defined lifestyle factors impacted by PD
Work Productivity and Activity Impairment | 4 months, 1 year, 2 years, 3 years
  Change in Work Productivity and Activity Impairment Questionnaire (WPAI) from baseline. The WPAI Questionnaire includes questions regarding impacts to work productivity due to PD symptoms.
PKG scores | 4 months, 1 year, 2 years, 3 years
  Proportion of enrolled subjects in PKG+ group who are either unable to be brought into the target range or unable to be brought to a BKS ≤26. A higher score represents more severe bradykinesia.

CONTACTS AND LOCATIONS:
Overall Officials: Raja Mehanna, MD, Principal Investigator — The University of Texas Health Science Center, Houston

REFERENCES:
- [Background] Pahwa R, Isaacson SH, Torres-Russotto D, Nahab FB, Lynch PM, Kotschet KE. Role of the Personal KinetiGraph in the routine clinical assessment of Parkinson's disease: recommendations from an expert panel. Expert Rev Neurother. 2018 Aug;18(8):669-680. doi: 10.1080/14737175.2018.1503948. Epub 2018 Jul 26. PMID 30032695
- [Background] Shulman LM, Gruber-Baldini AL, Anderson KE, Fishman PS, Reich SG, Weiner WJ. The clinically important difference on the unified Parkinson's disease rating scale. Arch Neurol. 2010 Jan;67(1):64-70. doi: 10.1001/archneurol.2009.295. PMID 20065131
- See also: Sponsor website — https://www.globalkineticscorporation.com/